CLINICAL TRIAL: NCT01174615
Title: Collection of Blood and/or Bone Marrow for Investigation and Characterization of Normal and Abnormal Cell Growth in Patients With Malignancy or Hematologic Disorders
Brief Title: Collection of Blood and/or Bone Marrow for Investigation and Characterization of Normal and Abnormal Cell Growth
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawing as this is not a clinical trial
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: UM200901
Record Dates: First submitted 2010-05-24; First posted 2010-08-03 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Leukemia
Keywords: Blood/bone marrow collection, hematologic diseases, leukemia
MeSH Terms: conditions — Leukemia; Hematologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue/cells from patients' samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
The collection of Blood and/or Bone Marrow from patients with blood disorders, blood cell malignancies and associated conditions will serve as a convenient and comprehensive source of tissue to give us further information about the differences between normal blood cells and blood cells of affected individuals. This will be an invaluable asset for understanding the biology of blood disorders. The collected samples will be used by investigators for studies including immunology, molecular biology and genetics to name a few.

ELIGIBILITY:
Inclusion Criteria:

* Selected patients over the age of 18 with hematologic malignancies or other blood disorders (leukemia, myeloproliferative disorders, lymphoma, other malignancies involving the bone marrow or patients with unexplained alterations in their complete blood count).

Patients who are scheduled to undergo a bone marrow aspirate and/or phlebotomy for other clinical indications will be asked to participate. They will be asked to donate an additional small aliquot of bone marrow and/or blood during the course of their already scheduled bone marrow aspiration or phlebotomy.

Exclusion Criteria:

* Patients with pre-existing medical conditions that might be exacerbated by the procedure of obtaining bone marrow or blood
* Patients who are allergic to Lidocaine, which is used as a local anesthetic, and who cannot receive a suitable substitute anesthetic.
* Patients who have a bleeding diathesis which might pose a problem with marrow aspiration.
* Patients unable to give informed consent.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 with blood and/or bone disorders (leukemia, myeloproliferative disorders, lymphoma etc.) with alterations of their blood counts.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2099-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
The study is designed to collect blood and bone marrow from patients with various hematological diseases. | On average, indefinite, or until death of participant
  The study is designed to collect blood and bone marrow from patients with various hematological diseases. The samples will be used for various research studies for better understanding of biology of various blood disorders including hematological malignancies. Relevant clinical and laboratory features and subsequent changes will be noted for correlation with these studies. The tissue/cells will be additionally banked and/or used for other investigations in the future.

SECONDARY OUTCOMES:
Collection of Blood and/or Bone Marrow for Investigation and Characterization of Normal and Abnormal Cell Growth in Patients With Malignancy or Hematologic Disorders | On average, indefinite, or until death of participant
  Develop a database of subjects who have donated samples for research as well as tissue banking, some of whom may be contacted again for consideration of additional studies in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Cerny, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States